CLINICAL TRIAL: NCT04146038
Title: Salsalate + Venetoclax/Decitabine for Patients With Acute Myelogenous Leukemia or Advanced Myelodysplasia/Myeloproliferative Disease
Brief Title: Salsalate, Venetoclax, and Decitabine or Azacitidine for the Treatment of Acute Myeloid Leukemia or Advanced Myelodysplasia/Myeloproliferative Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Professor of Medicine, Chief of Hematologic Malignancies Medical Oncology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 021905; NCI-2019-07031 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2019001209; Pro2019001209 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myeloblasts 10 Percent or More of Bone Marrow Nucleated Cells; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Azacitidine; Decitabine; Injections; salicylsalicylic acid; Sodium Salicylate; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (salsalate, decitabine, azacitidine, venetoclax) (Experimental): CYCLE 1: Patients receive salsalate PO BID until completion of cycle 1. 24-48 hours later or concurrent with salsalate, patients begin to receive decitabine IV for 10 days or azacitidine IV for 7 days. Starting 24 hour after salsalate, patients also receive venetoclax PO continuously until completion of cycle 1.
  CYCLE 2: Patients receive decitabine IV for 5 days or azacitidine IV for 7 days, salsalate PO BID, and venetoclax PO continuously.
  Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Decitabine; Drug: Salsalate; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Salsalate — Given PO
  Other Names: Disalcid; Mono-Gesic; o-Salicylsalicylic Acid; Salflex; Salicylsalicylic Acid; Salsitab
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the side effects of salsalate when added to venetoclax and decitabine or azacitidine in treating patients with acute myeloid leukemia or myelodysplasia/myeloproliferative disease that has spread to other places in the body (advanced). Drugs used in chemotherapy, such as salsalate, venetoclax, decitabine, and azacitidine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the tolerability of the addition of standard dose salsalate to the standard treatment combination of venetoclax + hypomethylating agent (HMA) (decitabine or azacitidine [5-azacytidine]).

SECONDARY OBJECTIVES:

I. Determine the remission rate and, when feasible, perform exploratory studies of:

Ia. Patterns of mutation clearance. Ib. Distribution of cells with low and high reactive oxygen species (ROS) content at various points during therapy.

OUTLINE:

CYCLE 1: Patients receive salsalate orally (PO) twice daily (BID) until completion of cycle 1. 24-48 hours later or concurrent with salsalate, patients begin to receive decitabine intravenously (IV) for 10 days or azacitidine IV for 7 days. Starting 24 hour after salsalate, patients also receive venetoclax PO continuously until completion of cycle 1.

CYCLE 2: Patients receive decitabine IV for 5 days or azacitidine IV for 7 days, salsalate PO BID, and venetoclax PO continuously.

Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven acute myelogenous leukemia (AML) or advanced myeloid malignancy [myelodysplasia; chronic myelomonocytic leukemia (CMML); or chronic myeloproliferative disease (MPD) each with >= 10% myeloblasts in blood or bone marrow]
* For patients with de novo AML: must not be a candidate for standard induction therapy based upon age, co-morbidities, patient choice, high risk features known to have poor outcomes with standard induction therapy (ELN high risk disease by cytogenetics, deoxyribonucleic acid [DNA] mutation profile or TP53 mutation)
* Patients with advanced myelodysplastic syndrome (MDS), secondary AML, relapsed/refractory AML, prior hypomethylating agent are eligible
* Patients must give informed consent
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional ULN
* Creatinine < 2 mg/dL

Exclusion Criteria:

* White blood cell (WBC) uncontrolled (> 15,000/uL) despite hydroxyurea or cytarabine x 3 days. Known central nervous system (CNS) AML
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient?s ability to complete the study, at the discretion of the investigator. Pregnant patients are excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Salsalate or other agents used in the study. Examples include aspirin
* The effects of venetoclax and decitabine or 5-azacytidine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 24 weeks after. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, therefore, known human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with treatment medications or other agents administered during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax): CYCLE 1: Patients receive salsalate by mouth daily ( PO BID) until completion of cycle 1. 24-48 hours later or concurrent with salsalate, patients begin to receive decitabine IV for 10 days or azacitidine IV for 7 days. Starting 24 hour after salsalate, patients also receive venetoclax PO continuously until completion of cycle 1.
  CYCLE 2: Patients receive decitabine IV for 5 days or azacitidine IV for 7 days, salsalate PO BID, and venetoclax PO continuously.
  Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given IV
  Decitabine: Given IV
  Salsalate: Given PO
  Venetoclax: Given PO
Period: Overall Study
Arm/Group | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax): CYCLE 1: Patients receive salsalate PO BID until completion of cycle 1. 24-48 hours later or concurrent with salsalate, patients begin to receive decitabine IV for 10 days or azacitidine IV for 7 days. Starting 24 hour after salsalate, patients also receive venetoclax PO continuously until completion of cycle 1.
  CYCLE 2: Patients receive decitabine IV for 5 days or azacitidine IV for 7 days, salsalate PO BID, and venetoclax PO continuously.
  Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given IV
  Decitabine: Given IV
  Salsalate: Given PO
  Venetoclax: Given PO
Arm/Group | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events Incidence With of Salicylate + Venetoclax + Decitabine
Description: Study drug associated adverse events during therapy
Time Frame: During the first 2 cycles, 56 days total
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax)
Number analyzed (Participants) | 5
Participants | 1

2. Secondary Outcome: Number of Participants With Complete or Partial Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: During the first 2 cycles 56 days total
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax)
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: During the first two cycles (56 days), up to 2 years
Arm/Group | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax)
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax) (N=5)
Febrile neutropenia (Infections and infestations) | 2 (4)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Salsalate, Decitabine, Azacitidine, Venetoclax) (N=5)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 (15)
Investigations (Investigations) | 5 (30)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (5)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (5)
Vascular disorders (Vascular disorders) | 2 (2)
Cardiac disorders (Cardiac disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 1 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT04146038/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT04146038/ICF_001.pdf